CLINICAL TRIAL: NCT00783172
Title: OGF & Gemcitabine: Novel Treatment for Pancreatic Cancer Phase I, A Safety and Toxicity Study
Brief Title: Opioid Growth Factor (OGF) and Gemcitabine: Novel Treatment for Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Problems with IRB
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSU-20978 and 35686EP; 1R03CA129581 (NIH)
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2013-02

CONDITIONS: Pancreatic Cancer
Keywords: pancreas; pancreatic cancer; cancer; Opioid Growth Factor; OGF; gemcitabine; chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Gemcitabine; Enkephalin, Methionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OGF & Gemcitabine (Experimental): Opioid Growth factor 250 ug/kg IV once a week. Gemcitabine 1000 mg/m2 weekly for 7 out of 8 weeks induction then every 3 out of 4 week cycles.
  Interventions: Drug: Gemcitabine; Biological: Opioid Growth Factor (OGF)

INTERVENTIONS:
Drug: Gemcitabine — 1000mg/m2, IV (in the vein) over 30 minutes after treatment with OGF; first cycle is consecutive seven weeks and one week off; subsequent cycles are three weeks on and one week off.
  Other Names: Gemzar
Biological: Opioid Growth Factor (OGF) — Initial treatment is 150ug/kg (based on body weight of the patient) in a volume of 50ml sterile saline, IV (in the vein) over 45 minutes; subsequent treatments at dose of 250ug/kg
  Other Names: [Met]5-enkephalin

SUMMARY:
It is hypothesized that OGF biotherapy may be safely administered in combination with gemcitabine to individuals with unresectable pancreatic cancer. The study includes two aims, the first is to evaluate the safety and toxicity of the combination of OGF and gemcitabine chemotherapy. The second aim of the trial is to study the efficacy of OGF and gemcitabine when used in combination.

DETAILED DESCRIPTION:
Pancreatic cancer is the 4th leading cause of cancer-related deaths in the United States with a median survival of 3-6 months and a five-year survival rate of 1% making it the worse of all gastrointestinal malignancies. The reason for the poor prognosis is related to failure to diagnose this cancer in early stages and the unresponsiveness of pancreatic cancer to conventional chemotherapy and radiation therapy. Gemcitabine has become the standard of care in treatment of advanced pancreatic cancer; however, the mean survival with gemcitabine is reported at only 5.6 months. Our research team has discovered a novel biotherapy called Opioid Growth Factor (OGF) that inhibits growth of pancreatic cancer in vitro, in animals, and in human subjects. A Phase 1 study with OGF has been completed and the maximum tolerated dose, safety and toxicity evaluated. Currently a Phase 2 trial is in progress to study the efficacy of OGF monotherapy in those who have not responded to standard treatment. Recent experiments from our basic science laboratories indicate a marked additive benefit in cancer inhibition when OGF is combined with gemcitabine. Additionally, animals receiving the combination regime were healthier than those treated with gemcitabine alone suggesting perhaps a protective effect of OGF to chemotherapy toxicity. It is hypothesized that OGF may be safely administered in combination with gemcitabine to individuals with unresectable pancreatic cancer. In order to test this hypothesis 22 eligible naïve patients with pancreatic cancer will be prospectively treated with standard doses of gemcitabine. Concomitantly, OGF will be administered weekly starting at 150 μg/kg and increasing to the Maximum tolerated dose of 250 μg/kg in order to determine the following specific aims: 1) evaluate the safety and toxicity of the combination of OGF biotherapy and gemcitabine; 2) determine whether the combination therapy alters the pharmacokinetics of either agent; and 3) study the efficacy of combination therapy on tumor size, patient survival, and time to progression of disease. The long-term goal of our research team involves translation of novel discoveries from the basic science laboratory into clinical practice with the ultimate goal of improving survival of patients with this devastating disease.

ELIGIBILITY:
Inclusion Criteria:

* unresectable and histological or cytological confirmation of adenocarcinoma of the pancreas and measurable disease by CT scan
* patient has not been previously treated for pancreatic cancer

Exclusion Criteria:

* history of cancer other than pancreatic cancer (excluding resected basal cell skin cancer or curative stage 1 cervical cancer if disease free for 5 years or more)
* previous treatment with chemotherapy for pancreatic cancer
* uncontrolled cardiovascular disease (congestive heart failure, symptoms of coronary artery disease, cardiac arrhythmias)
* suffered from myocardial infarction in preceding 6 months
* poorly controlled medical conditions including: asthma, chronic obstructive pulmonary disease, diabetes, seizure disorders, known brain metastases, hepatic or renal failure
* pregnant or nursing women
* known allergy to gemcitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-01; Primary Completion 2010-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
progression measured with CT scan | every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jill P Smith, MD, Principal Investigator — Penn State University
Locations (2):
- United States (2):
  - Lehigh Valley Hospital and Health Network, Allentown, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania

REFERENCES:
- [Background] Zagon IS, Jaglowski JR, Verderame MF, Smith JP, Leure-Dupree AE, McLaughlin PJ. Combination chemotherapy with gemcitabine and biotherapy with opioid growth factor (OGF) enhances the growth inhibition of pancreatic adenocarcinoma. Cancer Chemother Pharmacol. 2005 Nov;56(5):510-20. doi: 10.1007/s00280-005-1028-x. Epub 2005 Jun 10. PMID 15947928
- [Background] Smith JP, Conter RL, Bingaman SI, Harvey HA, Mauger DT, Ahmad M, Demers LM, Stanley WB, McLaughlin PJ, Zagon IS. Treatment of advanced pancreatic cancer with opioid growth factor: phase I. Anticancer Drugs. 2004 Mar;15(3):203-9. doi: 10.1097/00001813-200403000-00003. PMID 15014352
- [Background] Zagon IS, Smith JP, McLaughlin PJ. Human pancreatic cancer cell proliferation in tissue culture is tonically inhibited by opioid growth factor. Int J Oncol. 1999 Mar;14(3):577-84. doi: 10.3892/ijo.14.3.577. PMID 10024694
- [Background] Zagon IS, Hytrek SD, Smith JP, McLaughlin PJ. Opioid growth factor (OGF) inhibits human pancreatic cancer transplanted into nude mice. Cancer Lett. 1997 Jan 30;112(2):167-75. doi: 10.1016/s0304-3835(96)04566-1. PMID 9066724
- [Background] Smith JP, Bingaman SI, Mauger DT, Harvey HH, Demers LM, Zagon IS. Opioid growth factor improves clinical benefit and survival in patients with advanced pancreatic cancer. Open Access J Clin Trials. 2010 Mar 1;2010(2):37-48. doi: 10.2147/oajct.s8270. PMID 20890374
- See also: Penn State Hershey Clinical Trials Office — http://www.hmc.psu.edu/clinicaltrials/
- See also: Penn State Hershey General Clinical Research Center — http://www.hmc.psu.edu/gcrc/patientsvolunteers/index.html